CLINICAL TRIAL: NCT04345575
Title: Self-Administered Skills-Based Virtual Reality Intervention for Chronic Pain: A Randomized Controlled Pilot Study
Brief Title: Self-Administered Skills-Based Virtual Reality Intervention for Chronic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AppliedVR Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-03
Record Dates: First submitted 2020-03-31; First posted 2020-04-14 (Actual); Last update posted 2020-04-14 (Actual); Status verified 2020-04

CONDITIONS: Chronic Pain
Keywords: virtual reality; chronic pain; behavioral health; behavioral medicine
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Intervention Model Description: Parallel group design where enrolled participants are randomly assigned to one of two treatment groups: Virtual reality behavioral medicine for chronic pain or Audio behavioral medicine for chronic pain
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VR Group (Experimental): VR group participants were mailed an Oculus Go Virtual Reality headset preloaded with VR software developed by AppliedVR. Treatment content consisted of a variety of 21 sessions to support participants in learning cognitive and behavioral self-management skills based on evidence-based CBT principles and skills, biofeedback and mindfulness strategies used in pain management. The program was designed to improve self-regulation of cognitive, emotion, and physiological response to stress and pain.
  Interventions: Device: PainCare VR
- Audio Group (Active Comparator): The audio program consisted of the majority of the same narrative content contained in the VR program. Owing to VR having a visual and auditory media form, about one-third of the Audio program included didactic and experiential content that was not identifical but was closely matched to the VR content (sans references to visual imagery that would be confusing in the absence of visual content). Participants accessed 21 audio recordings on SoundCloud and asked to complete one session each day.
  Interventions: Other: Audio content

INTERVENTIONS:
Device: PainCare VR — Didactic content delivered in virtual reality to support participants in learning cognitive and behavioral self-management skills based on cognitive-based therapy, biofeedback, and mindfulness strategies for pain management.
  Arms: VR Group
Other: Audio content — The audio program consisted of the majority of the same narrative content contained in the VR program. Owing to VR having a visual and auditory media form, about one-third of the VR program could not be included in the audio. Participants accessed 21 audio recordings on SoundCloud and asked to complete one session each day.
  Arms: Audio Group

SUMMARY:
Chronic pain management is optimized with a multidisciplinary biopsychosocial treatment approach. However, patients have limited access to comprehensive care that includes behavioral medicine for chronic pain. Virtual reality (VR) is an immersive technology and emerging digital behavioral pain therapeutic with analgesic efficacy for acute pain. No scientific literature was found for skills-based VR behavioral programs for chronic pain populations.

The primary goal of this study was to evaluate the feasibility of a self-administered VR program that included content and skills informed by evidence-based cognitive behavioral treatment for chronic pain. The secondary goal was to determine the preliminary efficacy of the VR program in terms of average pain intensity and pain-related interference with activity, stress, mood, and sleep, and its impact on pain-related cognition and self-efficacy. The tertiary goal was to conduct a randomized controlled trial to compare the VR treatment to an audio-only treatment; this comparison isolated the immersive effects of the skills-based VR program, thereby informing potential mechanisms of effect.

DETAILED DESCRIPTION:
This randomized controlled clinical trial was conducted between March and May of 2019. Participants were recruited through online advertisements on Facebook and The Mighty, a digital health community. Screening included a 2-item measure to assess for anhedonia and depressive symptoms experienced over the past two weeks. Potential participants were excluded from the study if they endorsed experiencing either depression or anhedonia nearly every day, and the other more than half the days. Eligible study participants were English-fluent adults 18-65 years of age, with either self-reported chronic low back pain without radicular symptoms and/or fibromyalgia pain of > 6 months duration,[29] and with average pain intensity > 4 (using the 11-point Numerical Rating Scale; 0=no pain, 10=worst pain imaginable) over the past month at screening. Exclusionary criteria included cognitive impairment, medical condition predisposing one to nausea or dizziness, hypersensitivity to flashing light or motion, absence of stereoscopic vision, severe hearing impairment, facial/head injury that would cause discomfort with VR use, cancer-related pain, severe depression, active suicidality, and previous use of Pain Care VR.

After informed consent was obtained study participants were randomized one-to-one using a REDCAP Cloud random number generator and allocated to treatment group. All study procedures were completed remotely and no in-person visits were required. Study participants were not blinded to treatment group assignment due to the obvious nature of the mode of delivery of their assigned treatment. Participant compensation was prorated based on the number of surveys completed; participants received up to $30 in the form of an Amazon.com e-gift card following completion of the final study survey. The study was approved by the Western Institutional Review Board (Puyallup, WA).

Data collection consisted of electronically collected patient-reported measures and objective use data collected from the VR devices and audio access logs.

In accordance with the Initiative on Methods, Measurement, and Pain Assessment in Clinical Trials (IMMPACT) recommendations, multiple methods evaluated the importance of change in outcome measures across four recommended domains: pain intensity, health-related quality of life as defined by physical functioning, and ratings of overall Improvement.

Both treatment groups received the same didactic content delivered in distinct formats (VR vs. Audio). Treatment content consisted of a variety of sessions to support participants in learning cognitive and behavioral self-management skills based on evidence-based CBT principles and skills, biofeedback and mindfulness strategies used in pain management.

The 21-day program consisted of 4-8 treatment sessions from each content category with the duration of session length ranging from 1-15 minutes. Each treatment session was indexed as complete if participants initiated the experience. Participants were allowed to replay completed sessions.

ELIGIBILITY:
Inclusion Criteria:

* English-fluent
* adults 18-65 years old
* have either self-reported chronic low back pain without radicular symptoms and/or fibromyalgia pain of > 6 months duration
* average pain intensity > 4 (using the 11-point Numerical Rating Scale; 0=no pain, 10=worst pain imaginable) over the past month at screening.

Exclusion Criteria:

* Cognitive impairment
* Current or prior diagnosis of epilepsy, dementia, migraines or other neurological disease that may prevent the use of VR
* Hypersensitivity to flashing light or motion
* No stereoscopic vision or severe hearing impairment
* Injury to eyes, face or neck that prevents comfortable use of VR
* Pain related to cancer
* Active suicidal ideation or severe depression
* Previous use of Pain Care VR for pain

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-05-30 (Actual); Study Completion 2019-05-30 (Actual)

PRIMARY OUTCOMES:
VR use | Day 1 through Day 21
  VR use will be calculated as the total number of sessions launched for the VR group.
VR satisfaction | Day 22
  Participant satisfaction ratings will be assessed using the question, "How satisfied or dissatisfied are you with the ability of this VR (Audio) program to relieve your symptoms" on a 5-point scale (1=Extremely Dissatisfied to 5=Extremely Satisfied). Satisfaction with treatment will be reported as percentages for the satisfaction categories 1-5 (on day 22).
VR Nausea and motion sickness | Day 22
  Nausea and motion sickness will be assessed on day 22 (post-treatment survey) using the question, "Did you experience any motion sickness or nausea while using VR?" on 4-point with 0=Never, 1=Sometimes, 2=Often, and 3=Always. The proportion of participants who did not experience any nausea/motion sickness will be reported.

SECONDARY OUTCOMES:
Average Pain Intensity | Baseline and Day 21
  Compare between group (VR vs Audio) pre-post treatment pain intensity (0-10 numeric rating scale) end of treatment on Day 21.
Pain Interference | Baseline and Day 21
  Department of Defense/Veterans Administration (DoD/VA) Scale assesses pain interference over the previous 24 hours at two time points: Baseline and end of treatment on Day 21 (0=does not interfere; 10=completely interferes). Between group (VR vs Audio) pre-post treatment for pain interference will be compared.
Pain-related Activity Interference | Baseline and Day 21
  Department of Defense/Veterans Administration (DoD/VA) Scale assesses activity interference over the previous 24 hours at two time points: Baseline and end of treatment on Day 21 (0=does not interfere; 10=completely interferes). Between group (VR vs Audio) pre-post treatment for activity interference will be compared.
Pain-related Mood Interference | Baseline and Day 21
  Department of Defense/Veterans Administration (DoD/VA) Scale assesses mood interference over the previous 24 hours at two time points: Baseline end of treatment on Day 21(0=does not interfere; 10=completely interferes). The investigators will compare mood interference between group (VR vs Audio) pre-post treatment.
Pain-related Sleep Interference | Baseline and Day 21
  Department of Defense/Veterans Administration (DoD/VA) Scale assesses sleep interference over the previous 24 hours at two time points: Baseline end of treatment on Day 21 (0=does not interfere; 10=completely interferes). The investigators will compare sleep interference between group (VR vs Audio) pre-post treatment.
Pain-related Stress Interference | Baseline and Day 21
  Department of Defense/Veterans Administration (DoD/VA) Scale assesses stress interference over the previous 24 hours at two time points: Baseline end of treatment on Day 21 (0=does not interfere; 10=completely interferes). The investigators will compare stress interference between group (VR vs Audio) pre-post treatment .
Pain Catastrophizing | Baseline and Day 22
  Pain Catastrophizing Scale (PCS) assesses frequency of pain-related thoughts and feelings on a 0-4 scale (0=not at all; 4=all the time). The PCS is assessed at baseline and post-treatment at day 22. There is no specific time referent for this measure. The investigators compared PCS between group (VR vs Audio) pre-post treatment.
Pain Self-Efficacy | Baseline and Day 22
  The 2-item PSEQ (PSEQ-2) is used to assess pain self-efficacy. Respondents rate their responses to the items using a 7-point scale ranging from 0 (Not at all confident) to 4 (Completely confident). The two item scores are summed to create a total score. The investigators will compare pain self-efficacy (PSEQ-2) between group (VR vs Audio) pre-post treatment .

CONTACTS AND LOCATIONS:
Overall Officials: Beth Darnall, PhD, Principal Investigator — Stanford University
Locations (1):
- AppliedVR, Inc., Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Classification of chronic pain. Descriptions of chronic pain syndromes and definitions of pain terms. Prepared by the International Association for the Study of Pain, Subcommittee on Taxonomy. Pain Suppl. 1986;3:S1-226. No abstract available. PMID 3461421
- [Background] Turner JA, Anderson ML, Balderson BH, Cook AJ, Sherman KJ, Cherkin DC. Mindfulness-based stress reduction and cognitive behavioral therapy for chronic low back pain: similar effects on mindfulness, catastrophizing, self-efficacy, and acceptance in a randomized controlled trial. Pain. 2016 Nov;157(11):2434-2444. doi: 10.1097/j.pain.0000000000000635. PMID 27257859
- [Background] Cherkin DC, Sherman KJ, Balderson BH, Cook AJ, Anderson ML, Hawkes RJ, Hansen KE, Turner JA. Effect of Mindfulness-Based Stress Reduction vs Cognitive Behavioral Therapy or Usual Care on Back Pain and Functional Limitations in Adults With Chronic Low Back Pain: A Randomized Clinical Trial. JAMA. 2016 Mar 22-29;315(12):1240-9. doi: 10.1001/jama.2016.2323. PMID 27002445
- [Background] Williams AC, Eccleston C, Morley S. Psychological therapies for the management of chronic pain (excluding headache) in adults. Cochrane Database Syst Rev. 2012 Nov 14;11(11):CD007407. doi: 10.1002/14651858.CD007407.pub3. PMID 23152245
- [Background] Hughes LS, Clark J, Colclough JA, Dale E, McMillan D. Acceptance and Commitment Therapy (ACT) for Chronic Pain: A Systematic Review and Meta-Analyses. Clin J Pain. 2017 Jun;33(6):552-568. doi: 10.1097/AJP.0000000000000425. PMID 27479642
- [Background] Darnall BD. Psychological Treatment for Patients with Chronic Pain. Washington, D.C.: American Psychological Association Press; 2018.
- [Background] Darnall BD, Scheman J, Davin S, Burns JW, Murphy JL, Wilson AC, Kerns RD, Mackey SC. Pain Psychology: A Global Needs Assessment and National Call to Action. Pain Med. 2016 Feb;17(2):250-63. doi: 10.1093/pm/pnv095. Epub 2016 Jan 23. PMID 26803844
- [Background] Spiegel B, Fuller G, Lopez M, Dupuy T, Noah B, Howard A, Albert M, Tashjian V, Lam R, Ahn J, Dailey F, Rosen BT, Vrahas M, Little M, Garlich J, Dzubur E, IsHak W, Danovitch I. Virtual reality for management of pain in hospitalized patients: A randomized comparative effectiveness trial. PLoS One. 2019 Aug 14;14(8):e0219115. doi: 10.1371/journal.pone.0219115. eCollection 2019. PMID 31412029
- [Background] Hoffman HG, Richards T, Coda B, Richards A, Sharar SR. The illusion of presence in immersive virtual reality during an fMRI brain scan. Cyberpsychol Behav. 2003 Apr;6(2):127-31. doi: 10.1089/109493103321640310. PMID 12804024
- [Background] Gold JI, Belmont KA, Thomas DA. The neurobiology of virtual reality pain attenuation. Cyberpsychol Behav. 2007 Aug;10(4):536-44. doi: 10.1089/cpb.2007.9993. PMID 17711362
- [Background] Geenen R, Bijlsma JW. Deviations in the endocrine system and brain of patients with fibromyalgia: cause or consequence of pain and associated features? Ann N Y Acad Sci. 2010 Apr;1193:98-110. doi: 10.1111/j.1749-6632.2009.05290.x. PMID 20398014
- [Background] Nararro-Haro MV, Hoffman HG, Garcia-Palacios A, Sampaio M, Alhalabi W, Hall K, Linehan M. The Use of Virtual Reality to Facilitate Mindfulness Skills Training in Dialectical Behavioral Therapy for Borderline Personality Disorder: A Case Study. Front Psychol. 2016 Nov 2;7:1573. doi: 10.3389/fpsyg.2016.01573. eCollection 2016. PMID 27853437
- [Background] Parsons TD, Rizzo AA. Affective outcomes of virtual reality exposure therapy for anxiety and specific phobias: a meta-analysis. J Behav Ther Exp Psychiatry. 2008 Sep;39(3):250-61. doi: 10.1016/j.jbtep.2007.07.007. Epub 2007 Jul 25. PMID 17720136
- [Background] Parsons TD, Rizzo AA, Rogers S, York P. Virtual reality in paediatric rehabilitation: a review. Dev Neurorehabil. 2009 Aug;12(4):224-38. doi: 10.1080/17518420902991719. PMID 19842822
- [Background] Gold JI, Kim SH, Kant AJ, Joseph MH, Rizzo AS. Effectiveness of virtual reality for pediatric pain distraction during i.v. placement. Cyberpsychol Behav. 2006 Apr;9(2):207-12. doi: 10.1089/cpb.2006.9.207. PMID 16640481
- [Background] Atzori B, Lauro Grotto R, Giugni A, Calabro M, Alhalabi W, Hoffman HG. Virtual Reality Analgesia for Pediatric Dental Patients. Front Psychol. 2018 Nov 23;9:2265. doi: 10.3389/fpsyg.2018.02265. eCollection 2018. PMID 30532720
- [Background] Gold JI, Mahrer NE. Is Virtual Reality Ready for Prime Time in the Medical Space? A Randomized Control Trial of Pediatric Virtual Reality for Acute Procedural Pain Management. J Pediatr Psychol. 2018 Apr 1;43(3):266-275. doi: 10.1093/jpepsy/jsx129. PMID 29053848
- [Background] Atzori B, Hoffman HG, Vagnoli L, Patterson DR, Alhalabi W, Messeri A, Lauro Grotto R. Virtual Reality Analgesia During Venipuncture in Pediatric Patients With Onco-Hematological Diseases. Front Psychol. 2018 Dec 20;9:2508. doi: 10.3389/fpsyg.2018.02508. eCollection 2018. PMID 30618938
- [Background] Hoffman HG, Chambers GT, Meyer WJ 3rd, Arceneaux LL, Russell WJ, Seibel EJ, Richards TL, Sharar SR, Patterson DR. Virtual reality as an adjunctive non-pharmacologic analgesic for acute burn pain during medical procedures. Ann Behav Med. 2011 Apr;41(2):183-91. doi: 10.1007/s12160-010-9248-7. PMID 21264690
- [Background] Khadra C, Ballard A, Dery J, Paquin D, Fortin JS, Perreault I, Labbe DR, Hoffman HG, Bouchard S, LeMay S. Projector-based virtual reality dome environment for procedural pain and anxiety in young children with burn injuries: a pilot study. J Pain Res. 2018 Feb 14;11:343-353. doi: 10.2147/JPR.S151084. eCollection 2018. PMID 29491717
- [Background] Dascal J, Reid M, IsHak WW, Spiegel B, Recacho J, Rosen B, Danovitch I. Virtual Reality and Medical Inpatients: A Systematic Review of Randomized, Controlled Trials. Innov Clin Neurosci. 2017 Feb 1;14(1-2):14-21. eCollection 2017 Jan-Feb. PMID 28386517
- [Background] Sato K, Fukumori S, Matsusaki T, Maruo T, Ishikawa S, Nishie H, Takata K, Mizuhara H, Mizobuchi S, Nakatsuka H, Matsumi M, Gofuku A, Yokoyama M, Morita K. Nonimmersive virtual reality mirror visual feedback therapy and its application for the treatment of complex regional pain syndrome: an open-label pilot study. Pain Med. 2010 Apr;11(4):622-9. doi: 10.1111/j.1526-4637.2010.00819.x. Epub 2010 Mar 1. PMID 20202141
- [Background] Shiri S, Feintuch U, Weiss N, Pustilnik A, Geffen T, Kay B, Meiner Z, Berger I. A virtual reality system combined with biofeedback for treating pediatric chronic headache--a pilot study. Pain Med. 2013 May;14(5):621-7. doi: 10.1111/pme.12083. Epub 2013 May 9. PMID 23659372
- [Background] Garcia-Palacios A, Herrero R, Vizcaino Y, Belmonte MA, Castilla D, Molinari G, Banos RM, Botella C. Integrating virtual reality with activity management for the treatment of fibromyalgia: acceptability and preliminary efficacy. Clin J Pain. 2015 Jun;31(6):564-72. doi: 10.1097/AJP.0000000000000196. PMID 25551475
- [Background] Botella C, Garcia-Palacios A, Vizcaino Y, Herrero R, Banos RM, Belmonte MA. Virtual reality in the treatment of fibromyalgia: a pilot study. Cyberpsychol Behav Soc Netw. 2013 Mar;16(3):215-23. doi: 10.1089/cyber.2012.1572. PMID 23496678
- [Background] Wiederhold BK, Gao K, Sulea C, Wiederhold MD. Virtual reality as a distraction technique in chronic pain patients. Cyberpsychol Behav Soc Netw. 2014 Jun;17(6):346-52. doi: 10.1089/cyber.2014.0207. PMID 24892196
- [Background] Sulea C, Soomro A, Wiederhold BK, Wiederhold MD. Quantifying the effectiveness of virtual reality pain management: a pilot study. Stud Health Technol Inform. 2014;199:94-7. PMID 24875698
- [Background] Deyo RA, Dworkin SF, Amtmann D, Andersson G, Borenstein D, Carragee E, Carrino J, Chou R, Cook K, DeLitto A, Goertz C, Khalsa P, Loeser J, Mackey S, Panagis J, Rainville J, Tosteson T, Turk D, Von Korff M, Weiner DK. Report of the NIH Task Force on Research Standards for Chronic Low Back Pain. Int J Ther Massage Bodywork. 2015 Sep 1;8(3):16-33. doi: 10.3822/ijtmb.v8i3.295. eCollection 2015 Sep. PMID 26388962
- [Background] Dworkin RH, Turk DC, Farrar JT, Haythornthwaite JA, Jensen MP, Katz NP, Kerns RD, Stucki G, Allen RR, Bellamy N, Carr DB, Chandler J, Cowan P, Dionne R, Galer BS, Hertz S, Jadad AR, Kramer LD, Manning DC, Martin S, McCormick CG, McDermott MP, McGrath P, Quessy S, Rappaport BA, Robbins W, Robinson JP, Rothman M, Royal MA, Simon L, Stauffer JW, Stein W, Tollett J, Wernicke J, Witter J; IMMPACT. Core outcome measures for chronic pain clinical trials: IMMPACT recommendations. Pain. 2005 Jan;113(1-2):9-19. doi: 10.1016/j.pain.2004.09.012. No abstract available. PMID 15621359
- [Background] Turk DC, Dworkin RH, Burke LB, Gershon R, Rothman M, Scott J, Allen RR, Atkinson HJ, Chandler J, Cleeland C, Cowan P, Dimitrova R, Dionne R, Farrar JT, Haythornthwaite JA, Hertz S, Jadad AR, Jensen MP, Kellstein D, Kerns RD, Manning DC, Martin S, Max MB, McDermott MP, McGrath P, Moulin DE, Nurmikko T, Quessy S, Raja S, Rappaport BA, Rauschkolb C, Robinson JP, Royal MA, Simon L, Stauffer JW, Stucki G, Tollett J, von Stein T, Wallace MS, Wernicke J, White RE, Williams AC, Witter J, Wyrwich KW. Developing patient-reported outcome measures for pain clinical trials: IMMPACT recommendations. Pain. 2006 Dec 5;125(3):208-215. doi: 10.1016/j.pain.2006.09.028. Epub 2006 Oct 25. No abstract available. PMID 17069973
- [Background] Sullivan, M. J. L., Bishop, S. R., & Pivik, J. (1995). The Pain Catastrophizing Scale: Development and validation. Psychological Assessment, 7(4), 524-532. https://doi.org/10.1037/1040-3590.7.4.524
- [Background] Darnall BD, Sturgeon JA, Cook KF, Taub CJ, Roy A, Burns JW, Sullivan M, Mackey SC. Development and Validation of a Daily Pain Catastrophizing Scale. J Pain. 2017 Sep;18(9):1139-1149. doi: 10.1016/j.jpain.2017.05.003. Epub 2017 May 19. PMID 28528981
- [Background] Nicholas MK, McGuire BE, Asghari A. A 2-item short form of the Pain Self-efficacy Questionnaire: development and psychometric evaluation of PSEQ-2. J Pain. 2015 Feb;16(2):153-63. doi: 10.1016/j.jpain.2014.11.002. Epub 2014 Nov 14. PMID 25463701
- [Background] Dworkin RH, Turk DC, McDermott MP, Peirce-Sandner S, Burke LB, Cowan P, Farrar JT, Hertz S, Raja SN, Rappaport BA, Rauschkolb C, Sampaio C. Interpreting the clinical importance of group differences in chronic pain clinical trials: IMMPACT recommendations. Pain. 2009 Dec;146(3):238-244. doi: 10.1016/j.pain.2009.08.019. PMID 19836888
- [Background] Spiegel BM. Virtual medicine: how virtual reality is easing pain, calming nerves and improving health. Med J Aust. 2018 Sep 17;209(6):245-247. doi: 10.5694/mja17.00540. Epub 2018 May 21. No abstract available. PMID 29764343
- [Background] Darnall BD, Sturgeon JA, Kao MC, Hah JM, Mackey SC. From Catastrophizing to Recovery: a pilot study of a single-session treatment for pain catastrophizing. J Pain Res. 2014 Apr 25;7:219-26. doi: 10.2147/JPR.S62329. eCollection 2014. PMID 24851056